CLINICAL TRIAL: NCT00152542
Title: Follow up at School-age of Children Participating in the Nitric Oxide Ventilatory Approach (NOVA) Study
Brief Title: Follow-up at School-age of Children Who Participated in the Efficacy Study of Nitric Oxide for Premature Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 9549 (temp19); 29078
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2009-03

CONDITIONS: Prematurity, Respiratory Distress Syndrome,Hypoxemia
Keywords: Inhaled nitric oxide,; Lung recruitment,; Ventilatory approach,; Neurodevelopmental outcomes,; School age children
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled nitric oxide (Experimental)
  Interventions: Drug: Inhaled nitric oxide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled nitric oxide — 1 day of iNO at 10 ppm, then 5 ppm of iNO for days 2-7
  Arms: Inhaled nitric oxide
Drug: Placebo — No iNO given for days 1-7
  Arms: Placebo

SUMMARY:
Our previous data demonstrated that premature infants treated with inhaled nitric oxide at birth had improved neurodevelopmental outcomes at two years corrected age. We now wish to determine whether this benefit continues through school age.

DETAILED DESCRIPTION:
Two questionnaires (truncated versions of previously validated surveys), one for parent and another for teacher, for which written consent was previously obtained are being sent to parents. The teacher questionnaires will be delivered via parents. A clinic visit will accompany age appropriate neurodevelopmental examination, administration of the Functional Independence Measure for Children (WeeFIM) survey, and hearing and visual screening exams (if appropriate).

ELIGIBILITY:
Inclusion Criteria:

* Children who participated in NOVA study and are of school age

Exclusion Criteria:

* Children who participated in NOVA study but deceased post discharge

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Examine school-readiness at school-age in premature infants treated with iNO or placebo in the first week of life | 4-7 years of age (between 2005-2006)

SECONDARY OUTCOMES:
Examine health status at early school-age | 4-7 years of age (between 2005-2006)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Schreiber, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Comer Children's Hospital,, Chicago, Illinois, United States

REFERENCES:
- [Derived] Patrianakos-Hoobler AI, Marks JD, Msall ME, Huo D, Schreiber MD. Safety and efficacy of inhaled nitric oxide treatment for premature infants with respiratory distress syndrome: follow-up evaluation at early school age. Acta Paediatr. 2011 Apr;100(4):524-8. doi: 10.1111/j.1651-2227.2010.02077.x. Epub 2010 Dec 1. PMID 21054515